CLINICAL TRIAL: NCT02862093
Title: Transcranial Magnetic Stimulation in Alcohol Use Disorder: Effects on Dopamine Transporter and Alcohol Intake
Brief Title: Transcranial Magnetic Stimulation in Alcohol Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Giovanni Addolorato, Professor of Internal Medicine, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMSAlcoholDependeceStudy
Record Dates: First submitted 2016-08-03; First posted 2016-08-10 (Estimated); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deep rTMS (Active Comparator): The intervention consisted of deep rTMS of dorsolateral prefrontal cortex through the Brainsway Deep TMS System using an H-shaped coil . The motor threshold was measured by delivering a single pulse to the motor cortex. The site of stimulation was located 5.5 cm anterior to the point at which maximum stimulation of the abductor pollicis brevis muscle was reached. Each patient received a total of 12 rTMS sessions (three sessions per week): 20 trains per session at an intensity of 100% of the motor threshold, 50 pulses per train at a frequency of 10 Hertz, an inter-train interval of 15 seconds.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Placebo (Placebo Comparator): The sham stimulation consisted of rTMS sessions without an effective instrument operation.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Repetitive Transcranial Magnetic Stimulation of the dorsolateral prefrontal cortex

SUMMARY:
Repetitive Transcranial Magnetic Stimulation (rTMS) of the dorsolateral prefrontal cortex may affect neuro-adaptations associated with alcohol use disorder (AUD), potentially influencing craving and alcohol intake.

Investigators investigated alcohol intake and dopamine transporter (DAT) availability by Single Photon Emission Computed Tomography (SPECT) in the striatum of AUD patients before and after deep rTMS.

DETAILED DESCRIPTION:
The study included AUD patients. Patients were enrolled by the alcohol addiction unit of the Internal Medicine, Gastroenterology and Hepatology Department of the Catholic University in Rome, Italy, according to the inclusion criteria. Screening collection of medical history, physical, neurological and psychiatric examinations as well as laboratory tests were performed. Moreover, patients were underwent to baseline SPECT assessment of striatal DAT availability using 123I-N-ω-fluoropropyl-2β-carbomethoxy-3β-(4-iodophenyl) nortropane (123I-FP-CIT) as the radiotracer. Subsequently, patients were randomized in two groups (matched for gender and age) by a computer program for the REAL deep rTMS or SHAM. After weekly sessions of deep rTMS for four weeks, patients were underwent to the same clinical assessment as in the screening phase and second SPECT .

Moreover, the alcohol intake during both the four weeks prior to the enrollment and the 4 weeks of rTMS sessions were assessed through the Timeline Followback (TLFB) interview, an instrument providing a retrospective estimation of the number of drinks per drinking days, the number of drinking days, the number of abstinence days, the number of heavy drinking days and the total number of drinks. Patients were also evaluated with Alcohol Dependence Scale (ADS), Obsessive Compulsive Drinking Scale (OCDS), State-Trait Anxiety Inventory Scale (STAI Y1 and STAI Y2),Zung Self-Rating Depression Scale.

ELIGIBILITY:
Inclusion Criteria:

* At least two days a week of excessive alcohol consumption during the month prior to screening;
* Ability to provide informed consent;
* A Clinical Institute of Withdrawal Assessment in Alcohol Withdrawal score < 10;
* Willingness to abstain from or substantially reduce alcohol consumption;
* Permanent residence.

Exclusion Criteria:

* Clinically significant psychiatric diseases;
* Past or current abuse or dependence on substances other than alcohol or nicotine;
* Neurological disorders;
* Unstable medical conditions;
* Pacemakers, implanted metallic pumps, metal implant;
* History of complicated withdrawal symptoms;
* Current use of psychoactive drugs;
* Epilepsy;
* Current use of anticonvulsants, insulin or oral hypoglycemic agents;
* Positive urine toxicological screening;
* Pregnancy;
* Participation in other clinical trial in the last 60 days;
* Involvement in a compulsory medical treatment or pending criminal proceedings.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-01; Primary Completion 2013-02 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Dopamine Transporter availability in the striatum throgh Single Photon Emission Computed Tomography (SPECT) | Week 4

SECONDARY OUTCOMES:
Change From Baseline in alcohol intake | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Addolorato, Principal Investigator — Department of Internal Medicine, Catholic University of Rome, Italy
Locations (1):
- Catholic University of Rome, Rome, Rm, Italy